CLINICAL TRIAL: NCT04311346
Title: Cardiac MRI - Approaches for New Diagnostic Noninvasive Tools for the Detection of Cardiac Allograft Rejection
Brief Title: Cardiac MRI and Cardiac Allograft Rejection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tiina Ojala,MD, PhD, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: Helsinki UCH CMR
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Rejection Heart Transplant
Keywords: CMR; cardiac rejection; cardiac transplatation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac transplant: Patients exposed to cardiac transplantation
  Interventions: Diagnostic Test: Cardiac MR

INTERVENTIONS:
Diagnostic Test: Cardiac MR — Cardiac MR diagnostic tool for detection of acute rejection, double blind comparison with invasive cardiac biopsy

SUMMARY:
In this a prospective, blinded, collaboration study between pediatric and adult transplant departments. Cardiac MRI data on patient with heart transplantations will be collected during years 2020-2022. Based on sample size calculations, the data has enough power to answer the question, whether MRI can be used as a noninvasive diagnostic tool for detection of acute rejection as such or whether it can be used as fist line noninvasive screening tool for detecting those needing for the more detailed invasive study. A clinical protocol will be developed to optimize the management and outcome of the patients having cardiac transplantation aiming to decrease the number of invasive procedures in these patients.

DETAILED DESCRIPTION:
Background Heart transplantation is a treatment for select patients with end-stage heart failure. Improvements in immunosuppressive therapies and patient management have increased the life expectancy of heart transplant patients. One-year survivals are 90% and 80%, with 65 % and 49% of pediatric and adult patients surviving 8 - 15 years after transplantation in Finland, respectively. Despite this success, rejection remains the "Achilles heel" of heart transplantation. The early detection of acute rejection and cardiac allograft vasculopathy (chronic rejection) are paramount to avoiding graft loss. Unlike in kidney and liver transplantation, there are no clinically validated biomarkers for detecting heart transplant rejection.

Biopsy and invasive coronary angiography are widely accepted as the gold standard for diagnosing acute graft rejection and chronic rejection (vasculopathy) in both pediatric and adult heart transplant recipients, respectively. However, biopsies are invasive, and they carry a significant risk of complication regarding that majority of endocardial biopsies are performed in asymptomatic patients. In addition, the histologic assessment of biopsies is often subjective. Due to the lack of consensus, biopsy protocols are center-specific and depend on the experience and personal preference of the transplant team. Helsinki pediatric transplant protocol can be considered as high-intensity biopsy center. At best, the routine surveillance biopsies can detect late episodes of moderate to severe rejection in children with an 8% - 10% annual incidence up to 11 years after transplantation. However, there is no correlation between the intensity of biopsies and the incidence of rejection or 4-year mortality in the pediatric population, suggesting the need for other monitoring practices for rejection.

Cardiac MRI. Advanced multimodality imaging techniques, such as cardiac magnetic resonance imaging (MRI), may provide a future alternative to the monitoring practices for children and adults following heart transplantation. This has the potential to decrease the frequency of biopsies and radiation, especially in low-risk patients. Cardiac MRI can assess myocardial changes over time after transplantation. In heart transplant patients, MRI facilitates the detection of acute and chronic rejection and allows monitoring of gradual adverse remodeling. Volumetric assessment of the ventricles can further independently predict hospitalizations and mortality. The most widely investigated MRI parameters for detecting acute rejection are the T2 (indicates myocardial edema) and T1 relaxation times (indicates extracellular volume fraction (ECV) and fibrosis). Further, the assessment of global left ventricular function, myocardial strain analysis as well as late gadolinium enhancement (LGE) have been used for detection of chronic myocardial changes. Except for LGE and ECV, all of them can be measured noninvasively without the need for gadolinium contrast.

Even biopsy results may fail to predict rejection. A retrospective study of adults found that T2 time of ≥56 ms had a 97% negative predictive value for detecting acute rejection grade > 2. Interestingly, up to 80% of patients with a simultaneous negative biopsy but prolonged T2 relaxation time developed acute rejection in the next 30 days. The study suggested that T2 time measurement may be equal, or even superior to biopsy. However, the use of T2 relaxation time early after transplantation is limited, as it may be elevated in the first 25 days after transplantation regardless of the rejection status.

Contrast-enhanced MRI with gadolinium may provide additional information to T2 and T1 relaxation times and further limit the need for biopsies. It can identify areas of myocardial inflammation, scarring, and diffuse fibrosis, as well as assess myocardial perfusion. The prevalence of late gadolinium enhancement increases with the severity of rejection, whereas early gadolinium enhancement reflects extracellular space expansion secondary to acute necrosis and edema. Both myocardial edema (identified on T2- weighted imaging) and early myocardial contrast enhancement distinguish patients with International Society for Heart and Lung Transplantation (ISHLT) grade 2R rejection from those with grades 1R and 0R. Further, it has been reported that late enhancement in serially assessed transplant patients is associated with major adverse cardiac events and mortality. A recent study in 20 pediatric heart transplant patients showed that MRI-derived fibrosis markers correlate with the severity of fibrosis on biopsy. Although replacement fibrosis is irreversible, other MRI measurements change over time. Therefore, serial imaging can provide insight not only into disease progression but also on the efficacy of treatment. This is particularly relevant in acute rejection where the evaluation of myocardial edema with T2 mapping and interstitial expansion or fibrosis (T1 mapping ) can be accomplished with and without the administration of contrast agents and could easily limit the number of biopsies.

Hypothesis

Noninvasive cardiac MRI imaging can replace traditional invasive diagnostic procedures in detecting allograft rejection in cardiac transplant patients. This novel imaging strategy will reduce the cumulative stress and radiation and will guide clinical decision-making in these severely ill patients.

Patients and methods In this prospective blinded study, cardiac MRI data on new heart transplantations will be collected during years 2020-2021 (N = 72, including pediatric and adult patients). Estimated total count of invasive biopsies in the pediatric population is 100-150/2y samples, and the adult numbers will be three times higher (300-450/2y). The risk of the primary endpoint of acute rejection/immunoactivation is the highest during the first five years after transplantation. The immunoactivation occurs in 18 % and 10 % of samples taken <3 months and > 3 months after transplantation, respectively. Cardiac MRI immunoactivation/rejection findings will be blindly compared with the histological analysis of invasive endocardial biopsy done by one pathologist.

Sample size calculation (statistical consultation Tero Vahlberg, PhD): Clinically acceptable sensitivity for cardiac MRI to detect an acute rejection is 80%. Assuming an alpha level of 0.05, marginal error (precision) of 10% for sensitivity and 15% prevalence for rejection, the required total sample size is 410 samples. For specificity of 80% for cardiac MRI using the same assumptions, the required total sample size is 72 patients.

The required sample size is 410 biopsies and estimated time needed for data collection is two years. The data has then enough power to answer the question - whether MRI can be used as a noninvasive diagnostic tool for detection of acute rejection as such or whether it can be used as a fist line noninvasive screening tool for detecting those needing more detailed invasive study. MRI measurements published in adults for the detection of rejection or myocardial inflammation will be used. The detection of the secondary endpoint of vasculopathy/chronic rejection will be studied similarly to acute rejection. Cardiac MRI studies focusing on the vasculopathy findings will be carried out during the annual follow-up visits (two times during the study period/per patients, total n= 200). The MRI phenotype will be compared with invasive angiography findings. Advanced echocardiographic measurements will be further used for clinical, echocardiographic studies done in parallel with the cardiac MRI studies. The advanced echocardiographic methodology is based on the last 20 years research of group. Shortly, the methods to be used for functional MRI studies are the same as used in echo modality.

Ethical aspects The studies are designed to comply with the Helsinki Declaration and the Conventions of the Council of Europe on human rights. The results are reviewed and published anonymously. All clinical studies fulfill the general ethical requirements for clinical studies. The investigators have obtained following ethical permits from HUS ethical committee.

Clinical importance of the study Our project is realistic and timely. This project aims to promote noninvasive diagnostic strategies to replace traditional invasive procedures reducing cumulative stress and radiation in this group of severely ill heart transplant patients. This will be possible by creating a substantial amount of non-invasive research data on the myocardial mechanisms after transplantation. The investigators acknowledge that this project is ambitious. Our interdisciplinary research-group has vast experience of working with the proposed methods facilitating the success of this project. Our study results will build the foundations for new protocols to optimize the management and outcome of these patients. The methods the investigators use are validated, and the studies are well designed. The investigators are convinced that the results of the study will largely improve the clinical care of these patients. As MRI imaging is less expensive than invasive procedures, this approach will result in reduced health care costs in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cardiac Transplantation
* Patient must be suitable for cardiac CMR imagnining

Exclusion Criteria:

- Patient has pace maker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cardiac transplantations both in adults and in children have been centralized to Helsinki University Hospital, Finland. All patients both adults and children exposed to cardiac transplatations during the study period will be recruited to the study, if no contraindication for cardiac MR examination.
  Sample size calculation: the required total sample size is 72 patients
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2020-03-07 (Actual); Primary Completion 2022-03-07 (Estimated); Study Completion 2024-03-07 (Estimated)

PRIMARY OUTCOMES:
Cardiac rejection | Month 1
  Grade 0- Grade >2
Cardiac rejection | Month 2
  Grade 0- Grade >2
Cardiac rejection | Month 3
  Grade 0- Grade >2
Cardiac rejection | Month 4
  Grade 0- Grade >2
Cardiac rejection | Month 5
  Grade 0- Grade >2
Cardiac rejection | Month 6
  Grade 0- Grade >2
Cardiac rejection | Year 1
  Grade 0- Grade >2
Cardiac rejection | Year 2
  Grade 0- Grade >2

CONTACTS AND LOCATIONS:
Overall Officials: Tiina Ojala, MD, PhD, Principal Investigator — Helsinki University Hospital, Finland
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taipale MA, Pentikainen MO, Martelius LA, Mutka A, Kytola SI, Kankainen M, Peltonen JI, Syrjala SO, Lahtiharju AJI, Lommi JJ, Jahnukainen TJ, Lemstrom KB, Ojala TH. Cardiac magnetic resonance in heart transplant recipients: histological, clinical and cell-free DNA validation. Eur Heart J Cardiovasc Imaging. 2025 Jul 31;26(8):1420-1428. doi: 10.1093/ehjci/jeaf145. PMID 40384031